CLINICAL TRIAL: NCT01278017
Title: The Role of Short-course Ceftriaxone Therapy in the Treatment of Severe Nontyphoidal Salmonella Enterocolitis
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Chang Gung Memorial Hospital (Other)
Responsible Party: Tsai Ming-Han, Chang Gung Memorial Hospital
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: CMRPG290361
Record Dates: First submitted 2010-11-25; First posted 2011-01-17 (Estimated); Last update posted 2011-01-17 (Estimated); Status verified 2010-11

CONDITIONS: Diarrhea
Keywords: nontyphoidal salmonellae; enterocolitis; ceftriaxone
MeSH Terms: conditions — Diarrhea; Enterocolitis | interventions — Ceftriaxone

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- ceftriaxone (Experimental)
  Interventions: Drug: ceftriaxone

INTERVENTIONS:
Drug: ceftriaxone — ceftriaxone ,parenteral route, 50mg/kg/day divided twice
  Other Names: Rocephine

SUMMARY:
The purpose of the investigators study is to evaluate if short-course of ceftriaxone therapy could shorten the clinical courses of severe nontyphoidal Salmonella enterocolitis in children and the excretion of Salmonella in feces.

DETAILED DESCRIPTION:
Nontyphoidal salmonellae (NTS) is one of the most important pathogens of gastroenteritis in humans. Although most nontyphoidal Salmonella infections result in self-limited gastroenteritis, invasive infections such as bacteremia, meningitis or extraintestinal infection could also occur. Antimicrobial therapy is not recommended for routine treatment of nontyphoidal salmonellosis and effective antibiotic treatment is essential if NTS infection spreads beyond the intestine such as bacteremia, meningitis or osteomyelitis.

Although some reports revealed that antimicrobial therapy may be beneficial for shortening the clinical courses of severe NTS enterocolitis, most of them were based on clinical observations, not based on the results of objective examinations. Thus, the use of antibiotics in the treatment of patients with severe NTS gastroenteritis is still controversial in clinical practice.

As a third generation cephalosporin, ceftriaxone has a higher concentration than conventional antibiotics such as ampicillin and trimethoprim-sulfamethoxazole in the intestinal mucosa and gallbladder. Besides, ceftriaxone maintains relatively lower resistance rate in Salmonella than those of other conventional antibiotics. So the purpose of our study is to evaluate if short-course of ceftriaxone therapy could shorten the clinical courses of severe NTS enterocolitis in children and the excretion of Salmonella in feces. The investigators think that the study may be helpful for clinicians in the treatment of severe NTS enterocolitis in children, especially on the judgments of the choices and the treatment cures of antibiotics.

ELIGIBILITY:
Inclusion Criteria:

* Children with suspected severe Salmonella enterocolitis
* defined as those with a high fever (core body temperature ≥ 38.5℃) persisting for longer than 48 hours
* diarrhea with mucous and bloody-tinged stool.

Exclusion Criteria:

* Children with a toxic appearance, severe vomiting and abdominal distension
* suggestive of sepsis or toxic megacolon, those with an increased risk of invasive NTS diseases
* immunosuppressive illnesses
* had taken antibiotics during the 7 days before the visit will be excluded.

Ages: 3 Months to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 200 (Estimated)
Dates: Start 2010-08; Primary Completion 2011-06 (Estimated); Study Completion 2012-07 (Estimated)

PRIMARY OUTCOMES:
To evaluate if short-course of ceftriaxone therapy could shorten the clinical courses of severe NTS enterocolitis in children and the excretion of Salmonella in feces. | Three months
  Patients will be separated into 2 groups. One is treated with parenteral ceftriaxone and the other is treated with supportive drugs. Then we evaluate if short-course of ceftriaxone therapy could shorten the clinical courses of severe NTS enterocolitis in children and the excretion of Salmonella in feces.

SECONDARY OUTCOMES:
PCR detection will be used for Salmonella in stool samples. | Three month
  Patients will be randomly separated into 2 groups. One is treated with ceftriaxone and the other is treated with supportive drugs. Then we will evaluate if short-course of ceftriaxone therapy could shorten the clinical courses of severe NTS enterocolitis in children and the excretion of Salmonella in feces.

CONTACTS AND LOCATIONS:
Overall Officials: Ming_Han Tsai, MD, Principal Investigator — Chang Gung Memorial Hospital, Keelung, Taiwan
Locations (1):
- Chang Gung Memorial Hospital, Taoyuan District, Taiwan